CLINICAL TRIAL: NCT03018691
Title: A Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Trial to Assess the Safety and Efficacy of 0.3% and 1% OPA-15406 Ointments When Administered for 4 Weeks in Pediatric Patients With Atopic Dermatitis
Brief Title: Phase 2 Study of OPA-15406 Ointment in Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 271-102-00002; JapicCTI-173484 (Other: Japic)
Record Dates: First submitted 2017-01-06; First posted 2017-01-12 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.3% OPA-15406 Ointments (Experimental): Subjects were treated with assigned 0.3% OPA-15406 ointment twice daily.
  Interventions: Drug: OPA-15406
- 1% OPA-15406 Ointments (Experimental): Subjects were treated with assigned 1% OPA-15406 ointment twice daily.
  Interventions: Drug: OPA-15406
- Placebo Ointments (Placebo Comparator): Subjects were treated with assigned 0% OPA-15406 ointment twice daily.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: OPA-15406
  Arms: 0.3% OPA-15406 Ointments; 1% OPA-15406 Ointments
Drug: Placebos
  Arms: Placebo Ointments

SUMMARY:
To evaluate the safety, efficacy (dose response) and pharmacokinetics of 0.3% and 1% OPA-15406 when applied twice daily for 4 weeks in pediatric patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atopic dermatitis based on the criteria of Hanifin and Rajka

Exclusion Criteria:

* Subjects who have an atopic dermatitis or contact dermatitis flare-up defined as a sudden intensification of atopic dermatitis.
* Subjects who have an active viral skin infection.
* Subjects with a current or history of malignancy.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Ono, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (4):
- Japan (4):
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3% OPA-15406 Ointments: Subjects were treated with assigned 0.3% OPA-15406 ointment twice daily.
  OPA-15406
- 1% OPA-15406 Ointments: Subjects were treated with assigned 1% OPA-15406 ointment twice daily.
  OPA-15406
- Placebo Ointments: Subjects were treated with assigned 0% OPA-15406 ointment twice daily.
  Placebos
Period: Overall Study
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Started | 24 | 25 | 24
Completed | 22 | 24 | 17
Not Completed | 2 | 1 | 7
Not completed — Adverse Event | 1 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Withdrawal by parent/guardian | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments | Total
Number analyzed (Participants) | 24 | 25 | 24 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 25 | 24 | 73
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (3.8) | 7.9 (3.5) | 8.5 (3.1) | 8.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 5 | 21
  Male | 18 | 15 | 19 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese Subjects | 24 | 25 | 24 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 24 | 25 | 24 | 73

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Experiencing AEs
Description: The number of subjects experiencing AEs will be calculated for each treatment group.
  Treatment-emergent adverse events (TEAEs) occurring after the start of IMP administration are summarized. The number of subjects with events, the number of events is obtained for all the TEAEs reported.
Time Frame: Week 0-4
Measure: Number; unit: participants
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 24 | 25 | 24
participants | 11 | 14 | 12

2. Secondary Outcome: Responder Rate of Investigator's Global Assessment(IGA) of Disease Severity at Week4
Description: The investigator or subinvestigator assessed the skin symptoms using IGA. The investigator or subinvestigator scored the severity (0 = clear, 1 = almost clear, 2 =mild, 3 = moderate, 4 = severe/very severe) of the overall symptoms of the treatment area (erythema, infiltration, papules, effusion and scab formation) from baseline to Week4. Incidence of success in IGA was defined as the rate of subjects whose IGA score was 0 (clear) or 1 (almost clear) and had improved by at least 2 grades (responders) from baseline.
Time Frame: Baseline and Week 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 24 | 25 | 24
Percentage of participants | 37.50 [18.80 to 59.41] | 40.00 [21.13 to 61.33] | 8.33 [1.03 to 27.00]

3. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: The investigator or sub investigator assessed the symptoms of AD using EASI. EASI's minimum and maximum scores are 0 and 72 scores respectively. The higher the EASI score is, the more severe the symptoms of AD, and a negative change from the baseline means improvement and a positive change means worsening. The investigator or sub investigator scored the severity (0-3 points) and affected BSA (%) based on the 4 symptoms (erythema, infiltration/papules, excoriation, and lichenification) on the 4 body regions (face, neck and head ; upper limbs ;; and lower limbs). Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 23 | 24 | 18
score on a scale | -5.33 (1.28) | -5.52 (1.26) | 0.56 (1.36)

4. Secondary Outcome: Change From Baseline in Visual Analogue Scale(VAS) for Pruritus Score
Description: The investigator or subinvestigator evaluated the level of pruritus based on VAS. The subjects aged 7 to 14 years old marked the point of pruritus intensity during the last 24 hours on a 0 to 100mm VAS, with 0 being no pruritis to 100 being very severe pruritis.For subjects aged 2 to 6 years, this would not be evaluated. The negative value showed the degree of improvement.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: mm
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 16 | 16 | 14
mm | -18.00 (7.27) | -17.21 (7.29) | 8.19 (7.58)

5. Secondary Outcome: Change From Baseline in Verbal Rating Scale(VRS) for Pruritus Score
Description: The investigator or subinvestigator evaluated the pruritus intensity based on VRS. The subjects aged 7 to 14 years old evaluated the pruritus intensity according to the following criteria. The subjects recorded the level of pruritus and the time and date of evaluation in a pruritus diary.
  0 : None
  1. : Mild
  2. : Moderate
  3. : Severe For subjects aged 2 to 6 years, this would not be evaluated. The negative value showed the degree of improvement.
Time Frame: Baseline, Hour 156
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 15 | 17 | 14
score on a scale | -0.83 (0.18) | -0.73 (0.19) | 0.30 (0.11)

6. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure(POEM) Score
Description: The investigator or sub investigator evaluated eczema according to the POEM. The subjects answered 7 questions about their eczema by 0-4 points per question. The POEMS's minimum and maximum scores are 0 and 28 scores respectively. The higher the POEM score is, the more severe the symptoms are, and a negative change from the baseline means improvement and a positive change means worsening. If it is difficult for subjects to answer the questions, their parents answered them instead. Number of participants analyzed represents number of participants with data at both Baseline and Week4. Participants who have no data were excluded.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 23 | 24 | 18
score on a scale | -4.33 (1.16) | -4.37 (1.14) | 2.26 (1.24)

7. Secondary Outcome: Change From Baseline in Percentage Affected Body Surface Area
Description: The investigator or subinvestigator drew the affected BSA (range of skin eruption at the time of examination) on the human body drawing to determine the affected areas (%) on the respective 4 body regions (face, neck, and head; upper limbs; trunk; and lower limbs). One palm of the subject corresponds to 1% BSA. The negative value showed the degree of improvement.
Time Frame: Baseline, Week 8, 16, 24
Measure: Mean (Standard Error); unit: percentage of Affected Body Surface Area
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
Number analyzed (Participants) | 23 | 24 | 18
percentage of Affected Body Surface Area | -6.06 (2.36) | -8.21 (2.32) | 1.78 (2.53)

8. Secondary Outcome: Mean (SD) OPA-15406 Plasma Trough Concentrations at week1
Description: The plasma concentration of OPA-15406 was measured at Week 1. On the day of measurement, the subjects visited the trial site without morning Investigational Medicinal Product (IMP) administration.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.3% OPA-15406: Subjects were treated with assigned 0.3% OPA-15406 ointment twice daily.
- 1% OPA-15406: Subjects were treated with assigned 1% OPA-15406 ointment twice daily.
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 18 | 21
ng/mL | 0.842 (0.577) | 2.90 (2.74)

9. Secondary Outcome: Mean (SD) OPA-15406 Plasma Trough Concentrations at week4
Description: The plasma concentration of OPA-15406 was measured at Week 4. On the day of measurement, the subjects visited the trial site without morning Investigational Medicinal Product (IMP) administration.
Time Frame: week4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 20 | 22
ng/mL | 0.946 (1.16) | 2.21 (1.81)

10. Secondary Outcome: Mean (SD) Normalized OPA-15406 Plasma Trough Concentrations by Dose Derived From %BSA at week1
Description: The plasma concentration of OPA-15406 was measured at Week 1. On the day of measurement, the subjects visited the trial site without morning Investigational Medicinal Product (IMP) administration.Each plasma concentration was normalized by dose.
Time Frame: week1
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 18 | 21
ng/mL/mg | 0.196 (0.201) | 0.210 (0.174)

11. Secondary Outcome: Mean (SD) Normalized OPA-15406 Plasma Trough Concentrations by Dose Derived From %BSA at week4
Description: The plasma concentration of OPA-15406 was measured at Week 4. On the day of measurement, the subjects visited the trial site without morning Investigational Medicinal Product (IMP) administration.Each plasma concentration was normalized by dose.
Time Frame: week4
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | 0.3% OPA-15406 | 1% OPA-15406
Number analyzed (Participants) | 20 | 22
ng/mL/mg | 0.150 (0.111) | 0.166 (0.148)

ADVERSE EVENTS:
Time Frame: Treatment period
Arm/Group | 0.3% OPA-15406 Ointments | 1% OPA-15406 Ointments | Placebo Ointments
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 8/25 | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% OPA-15406 Ointments (N=24) | 1% OPA-15406 Ointments (N=25) | Placebo Ointments (N=24)
Influenza (Infections and infestations) | 2 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03018691/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT03018691/SAP_001.pdf